CLINICAL TRIAL: NCT05428670
Title: The Efficacy and Safety of ZR2 Versus R-CHOP-like Regimen for Elderly Patients With Newly Diagnosed Diffuse Large B Cell Lymphoma.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Haige Ye, Chief Physician, First Affiliated Hospital of Wenzhou Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HaigeYe
Record Dates: First submitted 2022-06-02; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Diffuse Large B Cell Lymphoma; Zanubrutinib; Elderly patients
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zanubrutinib+Rituximab+Lenalidomide (Experimental): The ZR2 regimen will be given from day 1 of each cycle of treatment. Each cycle will last for 21 days. Participants will receive a total of 6 cycles.
  Dosage:
  Zanubrutinib, 160 mg bid, po, day 2-21;
  Lenalidomide, 10-20 mg qd, po, day 2-14;
  Rituximab, 375 mg/m², ivgtt, day 1.
  Maintenance therapy:
  Patients who receive complete response or partial response after induction therapy will receive lenalidomide 10-20 mg qd po during 1-21 days in every 28 days, for a maximum of 2 years.
  Interventions: Drug: Zanubrutinib+Rituximab+Lenalidomide
- RCHOP/RCDOP (Active Comparator): The RCHOP/RCDOP regimen will be given from day 1 of each cycle of treatment. Each cycle will last for 21 days. Participants will receive a total of 6 cycles.
  Dosage:
  Rituximab, 375 mg/m², ivgtt, day 1;
  Cyclophosphamide, 500-750 mg/m², ivgtt, day 2;
  Doxorubicin, 50 mg/m², ivgtt day 2 (liposomal doxorubicin, 20-30 mg/m², ivgtt day 2 or Epirubicin, 50-60 mg/m², ivgtt day 2);
  Vincristine, 1.4 mg/m², iv day 2 or vindesine, 3mg/m², iv day 2;
  Prednisone, 100 mg qd, po day 2-6.
  Interventions: Drug: RCHOP/RCDOP

INTERVENTIONS:
Drug: Zanubrutinib+Rituximab+Lenalidomide — Zanubrutinib is a bruton' s tyrosine kinase inhibitor independently developed in China.
  Arms: Zanubrutinib+Rituximab+Lenalidomide
Drug: RCHOP/RCDOP — RCHOP/RCDOP is the classic treatment of diffuse large B cell lymphoma.
  Arms: RCHOP/RCDOP

SUMMARY:
This is a prospective, single-center, open-label clinical study designed to evaluate the efficacy and safety of the Zanubrutinib, Lenalidomide and Rituximab (ZR2) versus rituximab combined with CHOP or CDOP (R-CHOP or R-CDOP) in elderly patients with diffuse large B cell lymphoma treated for the first time.

DETAILED DESCRIPTION:
In this study, elderly DLBCL patients will be treated with ZR2 regimen for the first-line treatment. Investigators will compare the complete response rate, survival and incidence of adverse reactions between the RCHOP/RCDOP chemotherapy and the ZR2 regimen. In addition, immune function tests will be performed before treatment and every 2 courses after treatment, including peripheral blood lymphocyte-monocyte ratio, cytokines, immunoglobulins, T and B cells and their quantitative analysis. Patients with ZR2 regimen will undergo gene second-generation sequencing before treatment to compare the gene mutation differences between complete response (CR) and ≤ partial response (PR) in the efficacy of ZR2 regimen, in order to find biomarkers with better efficacy in ZR2 treatment. Moreover, investigators intend to conduct pharmacokinetics/pharmacodynamics (PK/PD) correlation analysis of ZR2 regimen and pharmacoeconomic evaluation of the two regimens.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed DLBCL
* Without treatment
* ≥ 65 years old
* Measurable lesions on CT or PET-CT before treatment
* Life expectancy of at least 3 months
* Voluntary participation with the consent of the patient
* Heart, kidney, liver and other organ function evaluation were basically normal before treatment

Exclusion Criteria:

* Patients who previously received chemotherapy
* Uncontrolled cardiovascular diseases, cerebrovascular diseases, thrombotic diseases, autoimmune diseases and serious infectious diseases
* Laboratory indicators before enrollment (unless caused by lymphoma):

  * Neutrophils < 1.5 × 10^9/L
  * Platelets < 80 × 10^9/L
  * Alanine aminotransferase or aspartate aminotransferase > 2 × ULN
  * Alkaline phosphatase or bilirubin > 1.5 × ULN
  * Creatinine > 1.5 × ULN
* Patients who cannot comply with the agreement due to mental diseases or other unknown reasons such as pregnancy and lactation
* HIV infection
* If HBsAg is positive, HBVDNA should be tested, and patients with positive DNA cannot be enrolled; if HBsAg is negative and HBcAb is positive (regardless of HBsAb status), HBVDNA should be tested, and patients with positive DNA cannot be enrolled
* Other uncontrolled medical conditions that may interfere with the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | At the end of Cycle 4 and Cycle 6 (each cycle is 21 days).
  Percentage of participants with complete response is determined on the basis of investigator assessments according to 2014 Lugano criteria.

SECONDARY OUTCOMES:
Overall survival | Baseline up to data cut-off (up to approximately 3 years).
  Overall survival is defined as the time from the date of randomization to the date of death from any cause.
Progression free survival | Baseline up to data cut-off (up to approximately 3 years).
  Progression-free survival is defined as the time from the date of randomization until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Incidence rate of adverse events | From enrollment to study completion, a maximum of 3 years.
  Percentage of participants with treatment-related adverse events is assessed by CTCAEv4.0.
Direct medical costs | At the end of Cycle 4 and Cycle 6 (each cycle is 21 days).
  Direct medical costs include personal expenses and medical insurance reimbursement expenses, mainly including examination expenses, disposal expenses, medical expenses, hospitalization expenses, and other expenses.
EQ-5D scores | At the end of Cycle 4 and Cycle 6 (each cycle is 21 days).
  EuroQoL (Quality of Life)-5 Dimensions (EQ-5D) is calculated for the pharmacoeconomics analysis to evaluate the quality of life in participants. EQ-5D is a participant answered questionnaire scoring 5 dimensions - mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The EQ-5D total score ranges from 0 (worst health state) to 1 (perfect health state) and 1 reflects the best outcome.
Maximum plasma concentration | The Cmax of zanubrutinib is determined at 2h postdose on day 2 of Cycle 2 (each cycle is 21 days) and the Cmax of lenalidomide is determined at 1h postdose on day 2 of Cycle 2 (each cycle is 21 days).
  Maximum plasma concentration (Cmax) is defined as maximum plasma concentration after dose.
Area under the plasma concentration-time curve | The AUC of zanubrutinib is determined at predose (0h), 2h and 24h postdose on day 2 of Cycle 2 (each cycle is 21 days) and the AUC of lenalidomide is determined at predose (0h), 1h and 24h postdose on day 2 of Cycle 2 (each cycle is 21 days).
  Area under the plasma concentration-time curve (AUC) is defined as the area under the curve from time zero to time of last quantifiable plasma concentration after dose.
Steady-state trough concentration | The Css,min of zanubrutinib is determined at 24h postdose on day 2 of Cycle 2 (each cycle is 21 days) and the Css,min of lenalidomide is determined at 24h postdose on day 2 of Cycle 2 (each cycle is 21 days).
  Steady-state trough concentration (Css,min) is defined as minimum plasma concentration after dose.

OTHER OUTCOMES:
cfDNA sequencing | Before treatment, at the end of Cycle 4 (each cycle is 21 days) and Cycle 6, and then every 6 months after the end of Cycle 6, a maximum of 2 years.
  Cell free deoxyribonucleic acid sequencing in peripheral blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No